CLINICAL TRIAL: NCT03323814
Title: Optimizing Peripheral Sensory Stimulation to Induce Sleep Slow Waves
Brief Title: Enhancing Sleep Slow Waves Using External Stimuli
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-0337 (H-2009-0052); A538900 (Other: UW Madison); SMPH\PSYCHIATRY\PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2016-04-12; First posted 2017-10-27 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Sleep, Slow-wave Sleep, Sleep Enhancement, Sleep Optimization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- short-sleepers: subset of participants will be recruited who report less than typical work/ weekday sleep in order to examine whether enhancing sleep with stimulation will reduce the amount of extra sleep subjects usually get on the weekends.
  Interventions: Device: Slow-wave optimization
- shift-workers: An additional subset of participants will be recruited who work evening shifts to see if enhanced sleep can counteract some of the effects of schedule shifting.
  Interventions: Device: Slow-wave optimization
- normal-sleepers: The first cohort will be used to optimize the the type and duration of sensory stimuli that will optimally enhance slow-waves.
  Interventions: Device: Slow-wave optimization

INTERVENTIONS:
Device: Slow-wave optimization — employing sensory stimulation to enhance slow waves
  Other Names: enhancing slow waves during non-rapid eye movement sleep

SUMMARY:
This is an observational study to determine if the presentation of sensory stimulation during sleep can increase slow-wave activity during non-rapid eye movement sleep

DETAILED DESCRIPTION:
This is a single-site,unblinded study at the University of Wisconsin to determine the effectiveness of various stimulation modalities and parameters to maximize effectiveness for increasing slow waves during both nocturnal sleep and during daytime naps The ongoing study is a necessary exploratory step towards the future development of non-pharmacological means to improve sleep by increasing SWA.

Several different stimulation modalities will be examined including: auditory (soft tones delivered to the subject through earphones); somatosensory (brief and painless electrical pulses delivered to the median nerve through electrodes placed at the wrist); vestibular (brief and painless electrical pulses delivered through electrodes placed near the mastoids); olfactory (light puffs of air, with or without mild odorants, delivered to the nostril(s) and/or mouth; visual (brief light flashes via strobe light). The amplitude (stimulus intensity) and frequency (number of stimuli per unit time) of stimulation presentation will be systematically varied to identify the ideal parameters for slow wave induction during sleep. For each stimulation modality and each subject, we will determine the range of stimulus intensity from the minimum level sufficient for perceptual response (e.g. - the lowest volume setting for an auditory stimulus that the subject can hear) to a stimulus level that the subject deems comfortable to still allow sleep. This is particularly important, as sleep maintenance during these experiments requires stimulus intensity low enough to avoid awakening the subject. Additionally, based on previous results from our laboratory, the effective range of stimulus intensity will vary substantially between subjects - both the identified range during wakefulness, as well as the range that induces slow waves but avoids waking during the sleep recording. Given this response variability, during the sleep recordings stimulus intensity will be adjusted, starting with the range determined in waking, to find the optimal intensity to inducing sleep slow waves (based on EEG response patterns), and avoiding subject awakening.

ELIGIBILITY:
Inclusion Criteria:Able to provide written informed consent prior to admission.

* Able to understand and speak English;
* Left or right-handed subjects may be included.
* Age of ≥18 years and ≤ 75;
* Able to understand and speak English;
* Left or right-handed subjects may be included.
* Age of ≥18 years and ≤ 75;

Exclusion Criteria:

* Subjects taking medications that could affect sleep patterns (based on self-report and review with a study clinician).
* Subjects who have had travel in the last 2 weeks or who intend to travel during the 4 experimental weeks (for at-home subjects) with time zone shifts >1h;
* The investigator anticipates that the subject will be unable to comply with the protocol.
* Individuals who self-report a current severe or chronic medical condition or sleep disorder that may affect sleep patterns (based on self-report and review with a study clinician).
* Individuals who self-report a history of recurrent seizures or epilepsy or family history of hereditary epilepsy or have a history of medical conditions that could increase the chance of seizures (e.g. stroke, aneurysm, brain surgery, structural brain lesion).
* Subjects who do report not being consistent in their daily use of alcohol, caffeine, or nicotine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 healthy volunteers will participatea)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Enhancing slow-wave sleep | 10 years
  increase slow-wave activity during non-rapid eye movement sleep

CONTACTS AND LOCATIONS:
Overall Officials: Guilio Tononi, MD, PhD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No